CLINICAL TRIAL: NCT01240226
Title: An Open-Label, 2-Part Study to Determine the Relative Bioavailability of a Tablet Formulation of GDC-0941 and the Effect of Ketoconazole on the Pharmacokinetics of the GDC-0941 Tablet
Brief Title: A Study to Determine the Relative Bioavailability of a Tablet Formulation of GDC-0941 and the Effect of Ketoconazole on the Pharmacokinetics of the GDC-0941 Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GDC4931g
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2012-07

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine; Ketoconazole

ARMS (2):
- A (Experimental)
  Interventions: Drug: GDC-0941; Drug: ketoconazole
- B (Experimental)
  Interventions: Drug: GDC-0941; Drug: ketoconazole

INTERVENTIONS:
Drug: GDC-0941 — Oral repeating dose
  Arms: A
Drug: GDC-0941 — Oral repeating dose
  Arms: B
Drug: ketoconazole — Oral repeating dose

SUMMARY:
This will be a single-center, open-label, randomized, 2-part study to determine the relative bioavailability of GDC-0941 capsule and market-image tablet formulations and the effect of ketoconazole on the pharmacokinetics of the GDC-0941 market-image tablet formulation.

ELIGIBILITY:
Inclusion Criteria

* Medically healthy as determined by the absence of clinically significant findings in the physical examination, medical history, vital sign measurements, clinical laboratory tests, or 12-lead electrocardiograms (ECGs)
* For female subjects: postmenopausal and without recent history of menorrhea, surgically sterile or using an effective method of contraception such as oral or transdermal contraceptives, double-barrier contraception, intrauterine device, depot progesterone, or implanted contraceptive devices, from Day -1 until 45 days after study drug completion/discharge; female subjects must have a negative pregnancy test at Screening and on Day -1
* For male subjects: sterile or a sterile sexual partner, or agreement to use 2 forms of medically acceptable methods of contraception, one of which is a barrier, and agreement not to donate sperm from Screening throughout the study period and for at least 3 months after the last dose of study drug.

Exclusion Criteria

* History of clinical manifestations of significant metabolic (including type 1 and 2 diabetes), hepatic, renal, hematological, pulmonary, cardiovascular, endocrine, gastrointestinal (including gastric or duodenal ulcers), urological, neurological, or psychiatric disease, or cancer
* History of inflammatory arthritis
* History of symptomatic hypotension
* History of severe physical injury, direct impact trauma, or neurological trauma within a specified timeframe prior to initiation of study treatment
* History of seizure disorders
* History of bipolar or major depressive disorder
* History of stomach or intestinal surgery or resection (except appendectomy, hernia repair, and cholecystectomy)
* History or presence of an abnormal ECG
* History of ventricular dysrhythmias or risk factors for ventricular dysrhythmias
* History of alcoholism, drug abuse, or drug addiction
* Use of any nicotine-containing or nicotine-replacement products within a specified timeframe prior to initiation of study treatment
* Use of medications capable of inhibiting hepatic enzymes within a specified timeframe prior to initiation of study treatment
* Participation in any other investigational drug study in which receipt of an investigational study drug occurred within a specified timeframe prior to initiation of study treatment
* Use of any prescription medications/products including monoamine oxidase inhibitors, thioridazine, pimozide, or antidepressants within a specified timeframe prior to initiation of study treatment (2 weeks for antibiotics) (except hormone-replacement therapy or 2 weeks use of narcotics for pain)
* Any vaccination or immunization within a specified timeframe prior to initiation of study treatment
* Routine use of PPIs or histamine H2-receptor antagonists, or any use of these drugs within a specified timeframe prior to initiation of study treatment
* Known hypersensitivity to ketoconazole or other azole antifungals
* Use of any over-the-counter, nonprescription preparations (including supplements, vitamins, minerals, phytotherapeutic/herbal/plant-derived preparations, tryptophans, and St. John's wort) within a specified timeframe prior to initiation of study treatment
* Use of alcohol-containing, grapefruit-containing, or caffeine-containing foods or beverages within a specified timeframe prior to initiation of study treatment
* Donated blood within within a specified timeframe prior to initiation of study treatment
* Received blood products within a specified timeframe prior to initiation of study treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Incidence, nature, and severity of adverse events | Through study completion or early study discontinuation
Pharmacokinetic parameters of GDC-0941 (total exposure, maximum and minimum plasma concentration) | Prior to and after GDC-0941 dosing

CONTACTS AND LOCATIONS:
Overall Officials: Scott Holden, M.D., Study Director — Genentech, Inc.
Locations (1):
- Investigational Site, Austin, Texas, United States